CLINICAL TRIAL: NCT06602531
Title: A Phase 1, First-in-human, Randomized, Observer-blind, Parallel Design, Controlled, Dose Level and Schedule-finding Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of a Self-Amplifying mRNA Pandemic Influenza Vaccine (ARCT-2304) When Administered to Healthy Adults
Brief Title: Safety and Immunogenicity Study of Self-Amplifying RNA Pandemic Influenza Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARCT-2304-01
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Influenza, Human
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Low dose of ARCT-2304, Schedule 1, Young Adults (Experimental): Low dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Mid dose of ARCT-2304, Schedule 1, Young Adults (Experimental): Mid dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- High dose of ARCT-2304, Schedule 1, Young Adults (Experimental): High dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Control, Schedule 1, Young Adults (Active Comparator): Control Vaccine (dose 1) and placebo (dose 2) administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: Comparator vaccine younger adult and saline placebo vaccine
  Interventions: Biological: Control vaccine younger adults; Other: Placebo Vaccine
- Low dose of ARCT-2304, Schedule 1, Older Adults (Experimental): Low dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Mid dose of ARCT-2304, Schedule 1, Older Adults (Experimental): Mid dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- High dose of ARCT-2304, Schedule 1, Older Adults (Experimental): High dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Control, Schedule 1, Older Adults (Active Comparator): Older Adults Control Vaccine (dose 1) and placebo (dose 2) administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 1 Investigational Vaccine: Comparator vaccine older adult and saline
  Interventions: Biological: Control vaccine older adults; Other: Placebo Vaccine
- Low dose of ARCT-2304, Schedule 2, Young Adults (Experimental): Low dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Mid dose of ARCT-2304, Schedule 2, Young Adults (Experimental): Mid dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- High dose of ARCT-2304, Schedule 2, Young Adults (Experimental): High dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Control, Schedule 2, Young Adults (Active Comparator): Young Adults Control Vaccine (dose 1) and placebo (dose 2) administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: Comparator vaccine younger adult and saline placebo vaccine
  Interventions: Biological: Control vaccine younger adults; Other: Placebo Vaccine
- Low dose of ARCT-2304, Schedule 2, Older Adults (Experimental): Low dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Mid dose of ARCT-2304, Schedule 2, Older Adults (Experimental): Mid dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- High dose of ARCT-2304, Schedule 2, Older Adults (Experimental): High dose of ARCT-2304 administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: ARCT-2304
  Interventions: Biological: ARCT-2304
- Control, Schedule 2, Older Adults (Active Comparator): Older Adults Control Vaccine (dose 1) and placebo (dose 2) administered through intramuscular injection in the deltoid muscle.
  Interventions: 2-dose regimen, schedule 2 Investigational Vaccine: Comparator vaccine older adult and saline placebo vaccine
  Interventions: Biological: Control vaccine older adults; Other: Placebo Vaccine

INTERVENTIONS:
Biological: ARCT-2304 — Each participant will receive 2-dose regimen intramuscular (IM) dose into the deltoid muscle.
  Other Names: Self-Amplifying mRNA pandemic Influenza vaccine
  Arms: High dose of ARCT-2304, Schedule 1, Older Adults; High dose of ARCT-2304, Schedule 1, Young Adults; High dose of ARCT-2304, Schedule 2, Older Adults; High dose of ARCT-2304, Schedule 2, Young Adults; Low dose of ARCT-2304, Schedule 1, Older Adults; Low dose of ARCT-2304, Schedule 1, Young Adults; Low dose of ARCT-2304, Schedule 2, Older Adults; Low dose of ARCT-2304, Schedule 2, Young Adults; Mid dose of ARCT-2304, Schedule 1, Older Adults; Mid dose of ARCT-2304, Schedule 1, Young Adults; Mid dose of ARCT-2304, Schedule 2, Older Adults; Mid dose of ARCT-2304, Schedule 2, Young Adults
Biological: Control vaccine younger adults — Each participant will receive one intramuscular (IM) dose into the deltoid muscle.
  Other Names: Influenza vaccine
  Arms: Control, Schedule 1, Young Adults; Control, Schedule 2, Young Adults
Biological: Control vaccine older adults — Each participant will receive one intramuscular (IM) dose into the deltoid muscle.
  Other Names: Influenza vaccine
  Arms: Control, Schedule 1, Older Adults; Control, Schedule 2, Older Adults
Other: Placebo Vaccine — Each participant will receive one intramuscular (IM) dose into the deltoid muscle.
  Other Names: saline
  Arms: Control, Schedule 1, Older Adults; Control, Schedule 1, Young Adults; Control, Schedule 2, Older Adults; Control, Schedule 2, Young Adults

SUMMARY:
The goal of this clinical trial is to evaluate the safety and immune responses of three different dose levels a self-amplifying RNA pandemic influenza vaccine (ARCT-2304) in adults. The key objectives of the study are:

* To evaluate safety and reactogenicity of different dose levels of the ARCT-2304 vaccine
* To describe the Immune responses of different dose levels of the ARCT-2304 vaccine as measured by hemagglutination inhibition (HAI) and neuraminidase enzyme-linked lectin (ELLA) antibody responses

Researchers will compare the results with licensed influenza vaccines to select the most optimal dose level and schedule for vaccine administration in terms of safety and immunogenicity for further development of the vaccine.

Participants will receive 2 doses of the ARCT-2304 vaccine or 1 dose of licensed influenza vaccine and 1 dose of placebo.

They will be asked:

* to complete a daily diary for 7 days after each vaccination, answering questions how they have been feeling on that day.
* to provide blood samples at each visit in the clinic
* to comply with all study visits and procedures (e.g., be available for planned telephone contacts and unscheduled clinic visits, if required)

DETAILED DESCRIPTION:
Phase 1, first-in-human, randomized, controlled, observer blind, dose level and schedule-finding study, to evaluate the safety, reactogenicity, and immunogenicity of a self-amplifying mRNA pandemic influenza (H5N1) vaccine (ARCT-2304) when administered as a 2-dose vaccination series to healthy adults in comparison with an inactivated influenza vaccine.

Study drug (ARCT-2304 or control) will be administered as a 2-dose vaccination series as an intramuscular (IM) injection. The study comprises two parts.

In Part 1, 120 participants (young adults) will be randomized to one of the three dose levels of the ARCT-2304 vaccine or control vaccine. Participants will be further randomized to one of the two different vaccination schedules.

In Part 2, 80 participants (older adults) will be randomized to one of the three dose levels of the ARCT-2304 vaccine or control vaccine. Participants will be further randomized to one of the two different vaccination schedules.

Investigational Vaccine: ARCT-2304

Control Vaccines: licensed influenza vaccines

ELIGIBILITY:
Main Inclusion Criteria:

* Individuals are male or female adults 18-80 years of age.
* Healthy participants or participants with pre-existing stable medical conditions.
* Individuals of childbearing potential must be willing to adhere to contraceptive requirements.

Main Exclusion Criteria:

* Individuals with acute medical conditions or febrile illness, including body temperature ≥100.4°F (≥38.0°C measured by any method) within 3 days prior to randomization.
* Individuals with a known history of severe hypersensitivity reactions, including anaphylaxis, or other significant adverse reactions to any mRNA vaccine, influenza vaccine, or excipients.
* Individuals with a history of myocarditis, pericarditis, myopericarditis, or cardiomyopathy.
* Individuals who received any influenza vaccine within 3 months prior to first vaccine administration or plan to receive an influenza vaccine during the study period.
* Individuals who have received mRNA vaccination within 60 days before the first vaccine administration.
* Individuals who have received or plan to receive an A/H5N1 influenza vaccine and/or individuals who had substantial exposure to or direct contact with poultry, wild birds, live cattle, or raw milk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting local Adverse Events | For 7 days following each study vaccination
  Solicited local AEs including injection site pain, erythema, and swelling
Percentage of participants reporting systemic Adverse Events | For 7 days following each study vaccination
  Solicited systemic AEs including fatigue, headache, myalgia, arthralgia, nausea, dizziness, chills, and fever
Percentage of participants reporting unsolicited Adverse Events | For 28 days following each study vaccination
  Spontaneously reported adverse events and as elicited by investigational site staff
Percentage of participants reporting laboratory or vital signs abnormalities | For 28 days following each study vaccination
  Abnormal clinically significant values
Percentage of participants reporting serious adverse events, medically attended adverse events, adverse events of special interest, and adverse events leading to early termination | For 28 days following each study vaccination
  Spontaneously reported adverse events and as elicited by investigational site staff
Serum hemagglutination inhibition (HAI) antibody levels against the HA glycoprotein | For 28 days following study second vaccination
  HAI antibody levels expressed as GMT, GMFRs, SCRs, and HAI titers
Serum neuraminidase enzyme-linked lectin (ELLA) assay antibody levels against the NA glycoproteins | For 28 days following study second vaccination
  ELLA antibody levels expressed as GMT, GMFRs, SCRs, and HAI titers

SECONDARY OUTCOMES:
Percentage of participants reporting serious adverse events, medically attended adverse events, adverse events of special interest, and adverse events leading to early termination | For 240 days following study vaccination
  Spontaneously reported adverse events and as elicited by investigational site staff
Serum hemagglutination inhibition (HAI) antibody levels against the HA glycoprotein | For 240 days following study vaccination
  HAI antibody levels expressed as GMT, GMFRs, SCRs and HAI titers
Serum neuraminidase enzyme-linked lectin (ELLA) assay antibody levels against the NA glycoproteins | For 240 days following study vaccination
  ELLA antibody levels expressed as GMT, GMFRs, SCRs and HAI titers
Serum neutralizing (MN) antibody levels against the HA glycoprotein | For 28 days following study second vaccination
  MN antibody levels expressed as GMT, GMFRs, SCRs, and MN titers

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Arcturus Therapeutics
Locations (4):
- United States (4):
  - Velocity Clinical Research, La Mesa, California
  - Velocity Clinical Research, San Bernardino, California
  - Tekton Research, Longmont, Colorado
  - CTI Clinical Research Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be made available to study investigators at this time.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT06602531/ICF_000.pdf